CLINICAL TRIAL: NCT00809679
Title: A Multicenter, Randomized, Double-Blind, Parallel, Placebo-Controlled, Pilot Analgesic Efficacy and Safety Study of T-62 in Subjects With Postherpetic Neuralgia
Brief Title: Analgesic Efficacy and Safety Study of T-62 in Subjects With Postherpetic Neuralgia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Some patients experienced asymptomatic, transient elevations in liver transaminases
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K862-08-2002
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Postherpetic Neuralgia
Keywords: Postherpetic neuralgia; Varicella Zoster; Shingles; Neuropathic pain; Analgesia; Pain
MeSH Terms: conditions — Neuralgia, Postherpetic; Herpes Zoster; Neuralgia; Agnosia; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- T-62 100 mg bid (Experimental)
  Interventions: Drug: T-62 Dose 1
- T-62 200 mg bid (Experimental)
  Interventions: Drug: T-62 Dose 2
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: T-62 Dose 1 — Capsule dosage form 100 mg bid
  Arms: T-62 100 mg bid
Drug: T-62 Dose 2 — Capsule dosage form 200 mg bid
  Arms: T-62 200 mg bid
Other: Placebo — Capsule dosage form placebo bid
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of T-62 in subjects with postherpetic neuralgia.

DETAILED DESCRIPTION:
Study K862-08-2002 is a multicenter, randomized, double-blind, placebo-controlled study assessing the analgesic efficacy and safety of T-62 in subjects with postherpetic neuralgia (PHN) and its associated pain. Up to 20 centers in the United States will participate in the trial. Two doses of T-62 and placebo will be evaluated in parallel design. Approximately 130 subjects will be enrolled to complete approximately 100 subjects. Each subject will complete a 7-day Screening Period , a 28-day Treatment Period, and a 14-day Post-Treatment Period. Each subject will complete 8 clinic visits over the course of the study during which procedures and assessments of safety, efficacy, and protocol compliance will be performed.

ELIGIBILITY:
Inclusion criteria (additional criteria apply):

1. Diagnosis of PHN made by primary treating physician and is experiencing pain for at least 3 months after the healing of a herpes zoster rash.
2. Subject is in general good health.
3. Females must be non-pregnant, non-lactating, and practicing an acceptable method of birth control or be surgically sterile or post-menopausal. Double barrier methods and abstinence are the only acceptable birth control methods for this study.

Exclusion Criteria (additional criteria apply):

1. Subject has a current acute disease or unstable chronic disease other than post herpetic neuralgia.
2. Subject has a clinically important history of a medical disorder (particularly cardiovascular, neurological [e.g., diabetic neuropathy], respiratory, or hepato-biliary systems [e.g., Gilbert Syndrome]) that would confound and/or interfere with the safety and efficacy evaluations defined in the protocol.
3. Subject is being treated for a medical condition that affects cardiac conduction.
4. Subject's plasma alanine aminotransferase (ALT) aspartate aminotransferase (AST), total bilirubin, and alkaline phosphatase (AP) values are not within the normal reference ranges.
5. Subject has a history of asthma requiring management for reactive airway disease in the last year.
6. Subject uses and is unwilling/unable to discontinue use of (A) Lyrica® (pregabalin), Cymbalta® (duloxetine), Neurontin® (gabapentin), topical lidocaine, topical capsaicin, or other medication specifically indicated (i.e., labeled) for the treatment of neuropathic pain, or (B) anticonvulsant medications to control post herpetic neuralgia.
7. Subject currently requires anticonvulsant medications to control seizures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Change in pain scores from baseline to following treatment. | weekly

SECONDARY OUTCOMES:
General safety monitoring (adverse reactions, vital signs, electrocardiograms, clinical laboratories) | weekly
Pharmacokinetics | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. Rolleri, Pharm. D., Study Director — King Pharmaceuticals is now a wholly owned subsidiary of Pfizer
Locations (13):
- United States (13):
  - Tucson, Arizona
  - Westlake Village, California
  - Bradenton, Florida
  - Naples, Florida
  - New Port Richey, Florida
  - Sunrise, Florida
  - Tampa, Florida
  - Lexington, Kentucky
  - Albuquerque, New Mexico
  - Winston-Salem, North Carolina
  - Oklahoma City, Oklahoma
  - San Antonio, Texas
  - Spokane, Washington